CLINICAL TRIAL: NCT02485535
Title: Phase I Study to Assess the Tolerability and Efficacy of Selinexor (KPT-330) as Single Agent to Eliminate Minimal Residual Disease and Maintain Remission in Patients With AML and High Risk MDS After Allogeneic Stem Cell Transplantation
Brief Title: Selinexor in Treating Patients With Intermediate- and High-Risk Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome After Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-1426; NCI-2015-00997 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-1426 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selinexor) (Experimental): Beginning on day 60-100 after allo-SCT without evidence of GVHD above grade 1 and disease relapse with stable hematopoietic recovery, patients receive selinexor PO on day 1 of each week or on days 1 and 3 of weeks 1-3. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selinexor

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330

SUMMARY:
This phase I trial studies the side effects and best dose of selinexor when given after stem cell transplant in treating patients with acute myeloid leukemia that is at intermediate or high risk of spreading or coming back (intermediate- or high-risk), or myelodysplastic syndrome that is at high risk of spreading or coming back (high-risk). Selinexor works to stop cancer growth by blocking an enzyme, which may cause cancer cells to die and also kill cells that cause the cancer to grow, which commonly do not respond to regular chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of selinexor in patients with hematologic malignancies, especially acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS), after allogeneic (allo)-stem cell transplant (SCT).

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of selinexor as maintenance treatment after allo-SCT.

II. To determine the incidence of non-relapse mortality. III. To determine 2 years post SCT progression-free survival (PFS) and overall survival rates.

IV. To determine the incidence of acute and chronic graft-versus-host disease (GVHD).

V. To assess lymphoid and myeloid chimerism post transplantation.

TERTIARY OBJECTIVES:

I. To analyze donor immune re-constitution after allo-SCT with selinexor maintenance.

II. To monitor minimal residual disease (MRD) by Wilms tumor 1 (WT1) polymerase chain reaction (PCR) during selinexor treatment in AML/MDS patients.

III. To characterize the physiopathology of the leukemia initiating cells (LIC) at the time of disease relapse on selinexor maintenance and compare that at initial diagnosis of the disease.

OUTLINE: This is a dose-escalation study.

Beginning on day 60-100 after allo-SCT without evidence of GVHD above grade 1 and disease relapse with stable hematopoietic recovery, patients receive selinexor orally (PO) on day 1 of each week or on days 1 and 3 of weeks 1-3. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent in accordance with federal, local, and institutional guidelines
* Patients underwent allo-SCT with intermediate risk and high risk AML and high risk MDS (defined by American Society for Blood and Marrow Transplantation [ASBMT] criteria), who are within 60 to 100 days after allo-SCT
* There is no evidence of disease relapse at the time of screening, and minimal residual disease (MRD) is acceptable
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count (ANC) > 1000 uL
* Platelets >= 20,000 without platelet transfusion
* Creatinine clearance > 30 cc/min calculated using the Cockcroft and Gault (1976) formula or measured
* Total bilirubin =< 2 mg/dl unless high indirect bilirubin is due to a congenital disorder
* Transaminases (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) =< 2.0 x upper limit of normal (ULN)
* Prothrombin time (PT) and partial thromboplastin time (PTT) =< 2 x ULN
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
* It is important patients understand the need to use birth control while on this study; female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening (< 3 days prior to first dose), male patients with partners of childbearing potential must agree to use effective contraception during the study period and a period of 3 months after the last dose of study drug; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose

Exclusion Criteria:

* Patients with acute GVHD grade II-IV
* Treatment with any investigational agent within three weeks prior to first dose in this study
* Major surgery within 2 weeks of first dose of study drug; patients must have recovered from the effects of any surgery performed greater than 2 weeks previously
* Patient has a concurrent active malignancy under treatment
* Unstable cardiovascular function:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or
  * Congestive heart failure (CHF) NYHA class >= 3, or
  * Myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable
* Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen)
* Known human immunodeficiency virus (HIV) infection
* Any medical condition which, in the investigator's opinion, could compromise the patient's safety
* Patients unable to swallow tablets or patients with malabsorption syndrome, or any other disease significantly affecting gastrointestinal function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
MTD of selinexor, determined according to incidence of DLT as graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 29 days

SECONDARY OUTCOMES:
Incidence of acute GVHD | Up to 2 years
  Summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented, as well as two-sided 95% CIs.
Incidence of adverse events (AEs), graded according to NCI CTCAE version 4.03 | Up to 2 years
  AEs will be summarized by patient incidence rates, therefore, in any tabulation, a patient contributes only once to the count for a given AE. The number and percentage of patients with any treatment emergent AE (TEAE) will be summarized for each treatment group, classified by system organ class and preferred term. The number and percentage of patients with TEAEs assessed by the investigator as at least possibly related to treatment will also be tabulated. The number and percentage of patients with any grade >= 3 TEAE will be tabulated in the same manner. Serious adverse events also tabulated.
Incidence of chronic GVHD | Up to 2 years
  Summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented, as well as two-sided 95% CIs.
Incidence of non-relapse mortality | Up to 2 years
  Summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented, as well as two-sided 95% confidence intervals (CIs).
Lymphoid and myeloid chimerism post transplantation | Up to 2 years
Overall survival (OS) | From the date of allo-SCT to the date of disease relapse or death, assessed up to 2 years
  The median duration of OS will be estimated based on the 50th percentile of the Kaplan-Meier distribution; additional summary statistics will be presented, including the 25th and 75th percentiles, 95% CIs on the median and other percentiles, and proportion of censored data. Kaplan-Meier survival rates will also be calculated. Additional exploratory Cox models may be used to determine the effect of other prognostic factors, such as MRD status at the time of treatment.
PFS | From the date of allo-SCT to the date of disease relapse or death, assessed up to 2 years
  The median duration of PFS will be estimated based on the 50th percentile of the Kaplan-Meier distribution; additional summary statistics will be presented, including the 25th and 75th percentiles, 95% CIs on the median and other percentiles, and proportion of censored data. Kaplan-Meier survival rates will also be calculated. Additional exploratory Cox models may be used to determine the effect of other prognostic factors, such as MRD status at the time of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States